CLINICAL TRIAL: NCT02330952
Title: Efficacy and Safety of Oral Corticosteroids for the Treatment of Acute Exacerbations of COPD in General Practice
Brief Title: Efficacy of Corticosteroids to Treat Outpatients With Acute Exacerbations of COPD
Acronym: BECOMEG
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AOM13195
Record Dates: First submitted 2015-01-01; First posted 2015-01-05 (Estimated); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Pulmonary Disease; Chronic Obstructive (MeSH)
Keywords: Double-blind method; Randomized Controlled trials
MeSH Terms: conditions — Lung Diseases | interventions — Prednisone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Prednisone (Experimental)
  Interventions: Drug: Prednisone
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Prednisone — 40mg/day per os for 5 days
  Arms: Prednisone
Drug: Placebo — 40mg/day per os for 5 days
  Arms: Placebo

SUMMARY:
Primary objective:

The aim of this study is to determine the efficacy and safety of five days of oral corticosteroids (40 mg / day) for the treatment of acute exacerbations of COPD (AECOPD) in outpatients.

DETAILED DESCRIPTION:
COPD is a major and growing public health issue. The vast majority of cases are cared for in primary care, both for follow-up in stable state and for treatment of exacerbations, which represent major events in the natural history of the disease.

Systemic corticosteroid treatment is often proposed for exacerbations treatment, although guidelines in this area are heterogeneous regarding precise indications of this treatment. The latest data from the literature, seems to show efficacy of oral corticosteroids but involved only patients seen at the hospital. General practitioners need evidence-base informations to choose whether or not they have to give oral corticosteroids to their patients ; therefore it is very important to better define the benefit-risk ratio and precise indications of oral corticosteroids as part of the care for COPD exacerbations.

The investigators built a randomized double-blind controlled trial to answer this question.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 40 years and over
* Smoking ≥ 10 pack-years
* Patients with suspected acute exacerbation of COPD
* Patients who gave their written informed consent to participate in the study

Exclusion Criteria:

* Known or suspected chronic respiratory disease other than COPD (asthma, bronchiectasis ...)
* Suspected pneumonia or pulmonary oedema
* Decision of hospitalization
* Patients taking oral corticosteroids running or stopped for less than a week before inclusion
* Pathology compromising compliance
* Fever unexplained by the current AECOPD
* Uncontrolled hypertension
* Uncontrolled diabetes
* Deep infectious disease
* History of ancient untreated tuberculosis
* Untreated peptic ulcer
* Unhealed wound
* Ulcerative Colitis
* Allergy to steroids
* Any severe or uncontrolled infections who are not specified as therapeutic indication in the SPC (Summary of Product Characteristics)
* Hepatitis, acute genital herpes, varicella, acute zoster
* Live attenuated vaccine, recent or planned
* Psychoses not controlled by treatment
* Hypersensitivity to prednisone or any of the excipients of Cortancyl®, including lactose intolerance
* Patients who have already been included in BECOMEG
* Patients who have to move within 8 weeks after inclusion in the study
* Patients who are not affiliated to the national health insurance

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 189 (Actual)
Dates: Start 2015-02-10 (Actual); Primary Completion 2017-05-23 (Actual); Study Completion 2017-05-23 (Actual)

PRIMARY OUTCOMES:
Treatment failure | 8 weeks
  Occurrence of one of the following events within 8 weeks after inclusion:
  * emergency visit (s) or consultation (s) (use of unscheduled care) related or not to the respiratory status of the patient
  * visit (s) to the emergency department, related or not to respiratory status
  * hospitalization (s), related or not to respiratory status
  * death, related or not to the respiratory status

SECONDARY OUTCOMES:
Quality of life-adjusted survival (Q-TWIST) | 8 weeks
  The Q-TWiST method (Quality-adjusted Time Without Symptoms or Toxicity) takes into account the survival times during which patients are asymptomatic and / or show signs of toxicity, affecting each of these periods a weighting coefficient between 0 (life without quality) and 1 (best possible quality of life).
MYMOP (Measure Yourself Medical Outcome Profile) | 8 weeks
  4 items assessed by the patient on a 7-level Likert scale from 1 (poor quality of life) to 7 (good quality of life)
COPD Assessment Test (CAT) | 8 weeks
  Questionnaire assessing the impact of COPD on quality of life
Dyspnea Medical Research Council (MRC) score | 8 weeks
  5-level dyspnea scale
Occurrence of each event | 8 weeks
  Rate of occurrence of each component of the primary endpoint within 8 weeks after inclusion
Treatment Failure related to respiratory status | 8 weeks
  Occurrence of one of the following events within 8 weeks after inclusion:
  * emergency visit (s) or consultation (s) (use of unscheduled care) related the respiratory status of the patient
  * visit (s) to the emergency department, related to respiratory status
  * hospitalization (s), related to respiratory status
  * death, related to the respiratory status
Self-managed relapse or recurrence | 8 weeks
  antibiotics and / or oral corticosteroids or other treatment taken after a consultation or on early prescription
Adverse events | 8 weeks
  All reported adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Christian Ghasarossian, MD, Principal Investigator — Département de Médecine Générale Faculté de Médecine Paris Descartes; Nicolas Roche, MD, PhD, Study Chair — Assistance Publique - Hôpitaux de Paris; Thomas Similowski, MD, PhD, Study Chair — Université Paris 6, Inserm, APHP; Jean-Laurent Thebault, MD, Study Chair — Département de Médecine Générale Faculté de Médecine Paris Descartes; Alain Lorenzo, MD, Study Chair — Département de Médecine Générale Faculté de Médecine Paris Descartes; François Bloede, MD, Study Chair — Département de Médecine Générale Faculté de Médecine Paris Descartes
Locations (1):
- Assistance Publique - Hopitaux Paris, Paris, France

REFERENCES:
- [Background] Thebault JL, Roche N, Abdoul H, Lorenzo A, Similowski T, Ghasarossian C. Efficacy and safety of oral corticosteroids to treat outpatients with acute exacerbations of COPD in primary care: a multicentre pragmatic randomised controlled study. ERJ Open Res. 2023 Sep 11;9(5):00057-2023. doi: 10.1183/23120541.00057-2023. eCollection 2023 Sep. PMID 37701369
- [Background] Rabbat A, Guetta A, Lorut C, Lefebvre A, Roche N, Huchon G. [Management of acute exacerbations of COPD]. Rev Mal Respir. 2010 Oct;27(8):939-53. doi: 10.1016/j.rmr.2010.08.003. French. PMID 20965408
- [Background] Thompson WH, Nielson CP, Carvalho P, Charan NB, Crowley JJ. Controlled trial of oral prednisone in outpatients with acute COPD exacerbation. Am J Respir Crit Care Med. 1996 Aug;154(2 Pt 1):407-12. doi: 10.1164/ajrccm.154.2.8756814.
- [Background] Walters JA, Wang W, Morley C, Soltani A, Wood-Baker R. Different durations of corticosteroid therapy for exacerbations of chronic obstructive pulmonary disease. Cochrane Database Syst Rev. 2011 Oct 5;(10):CD006897. doi: 10.1002/14651858.CD006897.pub2. PMID 21975757
- [Background] Walters JA, Gibson PG, Wood-Baker R, Hannay M, Walters EH. Systemic corticosteroids for acute exacerbations of chronic obstructive pulmonary disease. Cochrane Database Syst Rev. 2009 Jan 21;(1):CD001288. doi: 10.1002/14651858.CD001288.pub3. PMID 19160195
- [Background] Societe de Pneumologie de Langue Francaise. [Updated guidelines of the Societe de Pneumologie de Langue Francaise for the management of chronic obstructive pulmonary disease: essential points]. Rev Mal Respir. 2003 Apr;20(2 Pt 1):294-9. No abstract available. French. PMID 12844030